CLINICAL TRIAL: NCT06324812
Title: A Phase Ib/II Study to Evaluate the Safety, Pharmacokinetic and Efficacy of Recombinant Anti-interleukin-4 Receptor Alpha Monoclonal Antibody Injection (611) in Chinese Children and Adolescents (6 Years Old ≤ Age <18 Years Old) With Moderate to Severe Atopic Dermatitis
Brief Title: Evaluation of 611 in Chinese Children and Adolescents With Moderate to Severe Atopic Dermatitis
Status: Active, not recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Sunshine Guojian Pharmaceutical (Shanghai) Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SSGJ-611-PED-AD-Ib/II-01
Record Dates: First submitted 2024-03-14; First posted 2024-03-22 (Actual); Last update posted 2025-12-16 (Actual); Status verified 2025-07

CONDITIONS: Dermatitis, Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — entacapone

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 611 (Experimental): subcutaneous injection, 611 450/600mg (loading dose) + 300mg once every 2 weeks/4 weeks
  Interventions: Drug: Recombinant Anti-interleukin-4 Receptor Alpha Monoclonal Antibody Injection (611)

INTERVENTIONS:
Drug: Recombinant Anti-interleukin-4 Receptor Alpha Monoclonal Antibody Injection (611) — subcutaneous injection，611 450/600mg (loading dose) + 300mg once every 2 weeks/4 weeks

SUMMARY:
The primary objective of the study was to evaluate the safety and pharmacokinetic of 611 in Chinese children and adolescents with moderate to severe atopic dermatitis.

ELIGIBILITY:
Inclusion Criteria:

* Subjects or their legal guardians must be able to understand and comply with the study procedures. and must participate voluntarily and sign the written informed consent.
* When signing the informed consent form (ICF), Part 1: 12 years old ≤ age < 18 years old, weight ≥ 30kg; Part 2: 6 years old ≤ age < 12 years old, weight ≥ 15kg.
* AD (according to Hanifin-Rajka Criteria) that had been present for at least 1 years before the screening visit.
* (Investigator's Global Assessment) IGA ≥ 3 at screening and baseline visits.
* (Eczema Area and Severity Index) EASI ≥16 at screening and baseline visits.
* Participants with >=10 percent (%) body surface area (BSA) of AD involvement at screening and baseline visits.
* Baseline peak pruritus Numerical Rating Scale (NRS) average score for maximum itch intensity ≥4.
* With documented recent history (within 1 year before the baseline visit) of inadequate response to topical AD medication(s) or for whom topical treatments is medically inadvisable.
* Willing apply a stable dose of topical emollient (moisturizer) twice daily for at least the 7 consecutive days immediately before the baseline visit and continue for the duration of the study.
* Potentially fertile subjects (such as women who have had their first period or men who have had sperm implantation) must use highly effective contraception throughout the study period and for at least 3 months after the last dose.
* Patient, either alone or with help of parents/legal guardians, as appropriate, must be able to understand and complete study-related questionnaires.

Exclusion Criteria:

* Presence of skin comorbidities that may interfere with study assessments.
* Presence of active endoparasitic infections; or suspected endoparasitic.
* Any history of vernal keratoconjunctivitis (VKC) and atopic keratoconjunctivitis (AKC).
* History of malignancy within 5 years before the baseline visit.
* Participants who had a severe infection.
* Known or suspected history of immunosuppression.
* Active tuberculosis, unless that was well documented that the participants had adequately treated.
* Any medical condition that, in the opinion of the investigator, is serious or unstable and may affect the subject's safety and/or prevent the subject from completing the study.
* Treatment with topical drugs within 2 weeks before baseline; or systemic corticosteroids or immunosuppressive drugs within 4 weeks or 5 half-lives (whichever is longer) before baseline.
* Have been vaccinated with live (attenuated) vaccine within 4 weeks before baseline.
* The lab abnormalities at screening or baseline and not suitable for inclusion in the study judged by investigator.
* Patients who have active Hepatitis B, Hepatitis C or HIV infections as determined by positive results at Screening.
* History of alcohol or drug abuse within 6 months before baseline.
* History of hypersensitivity to 611 or their excipients.
* Have been participated in other clinical trials and used any experimental drugs within 8 weeks before baseline.
* Planned major surgical procedure during the patient's participation in this study.
* Patient is female who is pregnant, breastfeeding, or planning to become pregnant or breastfeed during the study.
* Any reason which, in the opinion of investigator, would prevent the subject from participating in the study.

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 124 (Estimated)
Dates: Start 2024-07-10 (Actual); Primary Completion 2026-08 (Estimated); Study Completion 2026-08 (Estimated)

PRIMARY OUTCOMES:
Adverse events (AEs), measurement of vital signs，physical examination，electrocardiogram and laboratory tests at each visit. | From baseline to week 24
  The incidence and severity of treatment emergent adverse event (TEAE), including Serious Adverse Event (SAE), as well as clinical symptoms, and any abnormalities of vital signs, physical examinations，electrocardiogram，laboratory tests and, etc.
Minimum concentration (Cmin) | From baseline to week 24
  Minimum concentration (Cmin) of 611

SECONDARY OUTCOMES:
Number of Participants with Eczema Area and Severity Index (EASI) - 75 Response (>= 75% Improvement in Score From Baseline) | From baseline to week 24
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Number of Participants with Investigator's Global Assessment (IGA) Score of "0" or "1" and Improvement From Baseline of Greater Than or Equal to (>=) 2 Points | From baseline to week 24
  The IGA is an assessment instrument used to rate the severity of AD globally based on a 5-point scale ranging from (0 = clear; 1 = almost clear; 2 = mild; 3 = moderate; 4 = severe), higher score indicated higher severity.
Number of Participants with Eczema Area and Severity Index (EASI) - 50 Response (>= 50% Improvement in Score From Baseline) | From baseline to week 24
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Number of Participants with Eczema Area and Severity Index (EASI) - 90 Response (>= 90% Improvement in Score From Baseline) | From baseline to week 24
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Number of Participants Who Achieved >=4 Points/ >=3 Points With Improvement From Baseline in Weekly Average of Pruritus Numerical Rating Scale (NRS) Score From Baseline | From baseline to week 24
  Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity.
Percentage Change From Baseline in EASI Score | From baseline to week 24
  The EASI score was used to measure the severity and extent of atopic dermatitis (AD) and measures erythema, infiltration, excoriation and lichenification on 4 anatomic regions of the body: head, trunk, upper and lower extremities. The total EASI score range from 0 (minimum) to 72 (maximum) points, with the higher scores reflecting the worse severity of AD.
Change From Baseline in Percent Body Surface Area (BSA) of AD Involvement | From baseline to week 24
  BSA affected by AD was assessed for each section of the body and reported as a percentage of all major body sections combined. The reported percentage of BSA was combined percentage of all major body sections，with the higher scores reflecting the worse severity of AD.
Change From Baseline in Weekly Average of Pruritus NRS | From baseline to week 24
  Pruritus NRS was an assessment tool that was used to report the intensity of a participant's pruritus (itch), during a 24-hour recall period. Participants were asked the following question: how would a participant rate his itch at the worst moment during the previous 24 hours (for maximum itch intensity on a scale of 0 - 10 [0 = no itch; 10 = worst itch imaginable]), higher scores indicated greater severity.
Change From Baseline in Children's Dermatology Life Quality Index (CDLQI) | From baseline to week 24
  CDLQI was a validated 10 question tool to measure the impact of skin disease on the quality of life (QOL) in children by assessing how much the skin problem has affected the participant over the past week. Nine questions were scored as follows: Very much = 3, Quite a lot = 2, Only a little = 1, Not at all or unanswered = 0. Question 7 has an added possible response, which was scored as 3. CDLQI equals the sum of the score of each question (maximum = 30, minimum = 0). Higher the score, the greater the impact on QOL.
Change From Baseline in Patient Oriented Eczema Measure (POEM) | From baseline to week 24
  POEM was a 7-item, validated questionnaire used to assess disease symptoms in children and adults. The format was a response to 7 items (dryness, itching, flaking, cracking, sleep loss, bleeding, and weeping) based on frequency of these disease symptoms during the past week (ie, 0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, and 4 = all days) with a scoring system of 0 to 28; the total score reflected the disease-related morbidity.

CONTACTS AND LOCATIONS:
Overall Officials: Lin Ma, MD, Principal Investigator — Beijing Children's Hospital
Locations (1):
- Beijing Children's Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: No